CLINICAL TRIAL: NCT03838263
Title: A Multicenter, Randomized, Open Label, Phase II Study Evaluating the Feasibility and Tolerance of Nivolumab Neoadjuvant Immunotherapy in High Risk HPV Driven Oropharynx Cancer
Brief Title: Feasibility and Tolerance of Nivolumab Neoadjuvant Immunotherapy in High Risk HPV Driven Oropharynx Cancer
Acronym: IMMUNEBOOST
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UNICANCER (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UC-0130/1804; 2018-000626-60 (EudraCT Number)
Record Dates: First submitted 2019-02-06; First posted 2019-02-12 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-02

CONDITIONS: Oropharynx Cancer
Keywords: Nivolumab; High-risk; HPV-driven oropharynx cancer
MeSH Terms: conditions — Oropharyngeal Neoplasms | interventions — Nivolumab; Chemoradiotherapy; Radiation; Cisplatin

STUDY DESIGN:
Intervention Model Description: In this study, there are 2 arms:
  * Experimental arm with nivolumab 2 infusions (2 weeks apart) before Standard of care chemoradiation for 7 weeks with high-dose cisplatin (100 mg/m²) at week 1, 4 and 7
  * Control arm: Standard of care chemoradiation for 7 weeks with high-dose cisplatin (100 mg/m²) at week 1, 4 and 7
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental arm (Experimental): Experimental arm with nivolumab 2 infusions (2 weeks apart) before Standard of care chemoradiation for 7 weeks with high-dose cisplatin (100 mg/m²) at week 1, 4 and 7
  Interventions: Drug: Nivolumab; Radiation: Chemoradiation
- Control arm (Active Comparator): Control arm: Standard of care chemoradiation for 7 weeks with high-dose cisplatin (100 mg/m²) at week 1, 4 and 7
  Interventions: Radiation: Chemoradiation

INTERVENTIONS:
Drug: Nivolumab — 2 nivolumab infusion (240 mg IV) 2 weeks apart (on day 1 and day 15) followed by standard chemoradiation.
  Other Names: ANY
  Arms: Experimental arm
Radiation: Chemoradiation — Standard of Care chemoradiation for 7 weeks (70 Gray delivered to the tumor by IMRT) with high-dose cisplatin (100mg/m2) at week 1, 4 and 7
  Other Names: Radiation + cisplatin

SUMMARY:
The aim of this research is to study the feasibility of neoadjuvant treatment before chemoradiation in "high risk" HPV-driven Oropharynx cancer

DETAILED DESCRIPTION:
Methodology:

Patient screened wil be randomized 2:1 between 2 arms:

* Experimental arm: Nivolumab 2 infusions (2 weeks part) before standard of care chemoradiation for 7 weeks with cisplatin at week 1, 4, and 7
* Control arm: Standard of care chemoradiation for 7 weeks with cisplatin at week 1, 4, and 7

Primary Objective:

To assess the feasibility and tolerance of neoadjuvant nivolumab treatment before chemoradiation in "high-risk" HPV-driven Oropharynx Cancer

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old
2. Histologically confirmed HPV-positive Oropharyngeal squamous cell carcinoma (OPSCC) amenable to curative treatment with RT-CT (HPV status is defined on the basis of the combination of 2 assays: p16 protein overexpression assessed by immunohistochemistry (IHC) and high-risk HPV DNA identification by in-situ Hybridization (ISH) or PCR. An HPV-driven OPSCC is defined as a tumor that is positive for both p16 IHC and HPV-DNA ISH or PCR)
3. According to the 8th TNM edition, eligible stages are as follow:

   * Irrespective of tobacco consumption: Stage T4 (any N), N2 or N3 (any T)
   * Only if tobacco consumption ≥10 pack- years: T1-3N1 and T3N0 (T1N0 and T2N0 irrespective of tobacco consumption are not eligible for the study)
4. Planned date of chemoradiation allowing 2 treatment infusions, 2 weeks apart
5. Eastern Cooperative Oncology Group (ECOG) performance status ≤1
6. Screening laboratory values must meet the following criteria (using CTCAE v5.0) and should be obtained within 7 days prior to the randomisation:

   1. Polynuclear neutrophils ≥1.5 x 10⁹/L
   2. Platelets ≥100 x 10⁹/L
   3. Hemoglobin ≥9.0 g/dL
   4. Alanine aminotransferase (ALAT)/aspartate transaminase (ASAT) ≤2.5 x upper limit of normal (ULN)
   5. Total Bilirubin ≤1.5 x ULN (except Gilbert Syndrome : <3.0 mg/dL)
   6. Creatinine clearance ≥60 mL/min (measured or calculated by Cockcroft and Gault formula)
7. Potentially reproductive patients must agree to use a highly effective contraceptive method while on treatment and up to 6 months after the end of chemoradiation
8. Women of childbearing potential must have a negative serum or urine pregnancy test done within 72 hours before randomisation
9. Patients must be willing and able to comply with scheduled visits, treatment plan, laboratory tests and other study procedures (including mandatory study-specific biopsies)
10. Subjects must have at least one lesion amenable to biopsy
11. Subjects must have at least one measurable lesion (different from the lesion amenable to biopsy) as per RECIST v1.1 to assess efficacy
12. Consent to provide archived tumour tissue sample, if available
13. Patients must be affiliated to a Social Security System
14. Patient information and written informed consent form signed

Exclusion Criteria:

1. Prior treatment for OPSCC
2. Prior treatment with anti PD-1/PD-L1 and CTLA-4
3. Distant metastases
4. Tumour embolization within 28 days prior to the first dose of study drug.
5. Contra-indication(s) to receive high-dose cisplatin as listed in the most updated Summary of Product Characteristics (including creatinine clearance <60 mL/min, pre-existing hearing loss or neurological disorder)
6. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, active peptic ulcer disease or gastritis, or psychiatric illness and social situations that would limit compliance with study requirement or compromise the ability of the subject to give written informed consent
7. Current or prior use of immunosuppressive medication within 14 days before the first dose, including intranasal and inhaled corticosteroids or systemic corticosteroids
8. Active or prior documented autoimmune or inflammatory disease within the 2 years prior to start of treatment (including inflammatory bowel disease [e.g., ulcerative colitis, Crohn's disease], celiac disease, irritable bowel disease, or other serious chronic gastrointestinal conditions associated with diarrhea; systemic lupus erythematosus; Wegener syndrome [granulomatosis with polyangiitis]; myasthenia gravis; Graves' disease; rheumatoid arthritis; hypophysitis, uveitis, etc.) The following are exceptions to these criteria:a) Subjects with vitiligo or alopecia, b) Subjects with hypothyroidism (e.g.,Hashimoto syndrome) stable on hormone replacement and c) Subjects with psoriasis not requiring systemic treatment (within the past 2 years)
9. History of primary immunodeficiency or organ transplant requiring immunosuppressive drugs
10. Patients with a known HIV, active hepatitis B or C infection
11. Other invasive malignancy within 3 years except for noninvasive malignancies such as cervical carcinoma in situ, non-melanomatous carcinoma of the skin or ductal carcinoma in situ of the breast that has/have been surgically cured
12. Pregnant women or women who are breast-feeding
13. Patients with any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the study
14. Individuals deprived of liberty or placed under the authority of a tutor
15. Severe infection requiring parenteral antibiotics treatment
16. Known history or active symptomatic interstitial lung disease
17. Patients with major surgery within 28 days, or open biopsy within 7 days, prior to randomisation. Patients must have recovered from major side effects of the surgery before randomisation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2019-07-25 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2024-11-20 (Actual)

PRIMARY OUTCOMES:
The rate of patients that fulfill the 3 or 5 conditions as described below (Feasibility assessment of nivolumab neoadjuvant treatment before chemoradiation) | Between baseline and until 3 months (at the end of chemoradiation)
  the rate of patients :
  (1) who can receive the 2 nivolumab infusions planned at D1 and between D14 to D16 among patients in the experimental arm And (2) who can receive chemoradiation at D30 (-2 /+7) after the second nivolumab infusion, without delay of more than 7 days with respect to the planned start of chemoradiation (RT-CT) among patients in the experimental arm And (3) with no radiotherapy break of one week or more, among patients in the experimental arm and patients in the control arm separately And (4) with minimal dose of radiotherapy (dose received >95% of theoretical dose) among patients in the experimental arm and patients in the control arm separately And (5) with minimal dose of chemotherapy of ≥200 mg/m² of cisplatin (CDDP) among patients in the experimental arm and patients in the control arm separately

SECONDARY OUTCOMES:
The incidence of Adverse Events related or not related to chemoradiation and Nivolumab | During treatment phase and until 90 days after the last fraction of radiotherapy
  Acute and delayed toxicities assessed according to national cancer institute (NCI) common terminology criteria for adverse events (CTCAE) version 5.0
Objective Response Rate in the experimental arm | Between baseline and up to 17 days after the second infusion of nivolumab
  Radiological response will be assessed according to RECIST 1.1.
Tumor Response in both arms | Between baseline and 3 months after the end of chemoradiation
  Radiological response will be assessed according to RECIST 1.1.
Overall Survival (OS) | Between baseline and 2 years after the end of chemoradiation
  the time from randomization to death from any cause
Locoregional control (LRC) | Between baseline and 2 years after the end of chemoradiation
  the absence of disease progression (radiological progression according to RECIST 1.1 or clinical progression) or recurrence at the site of the primary tumor and loco-regional lymph nodes.
Progression-Free Survival (PFS) | Between baseline and 2 years after the end of chemoradiation
  The time from randomization to progression or death from any cause
Objective Response Rate in the experimental arm | Between baseline and up to 17 days after the second infusion of nivolumab
  Standardized uptake value (SUV) evolution will be assessed by positron emission tomography (PET)-scan.
Tumor Response in both arms | Between baseline and 3 months after the end of chemoradiation
  SUV evolution will be assessed by PET-scan.

CONTACTS AND LOCATIONS:
Overall Officials: Haïtham MIRGHANI, MD, PhD, Principal Investigator — HOPITAL EUROPEEN GEORGES POMPIDOU
Locations (11):
- France (11):
  - Institut Sainte Catherine, Avignon
  - Hopital Beaujon, Clichy
  - Centre Léon Bérard, Lyon
  - Centre Antoine Lacassagne, Nice
  - Institut Curie, Paris
  - Hopital Europeen Georges Pompidou, Paris
  - Hopital Tenon, Paris
  - Centre Henri Becquerel, Rouen
  - Hopital Foch, Suresnes
  - Institut de cancerologie de Lorraine Alexis Vautrin, Vandœuvre-lès-Nancy
  - Institut Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: Yes
Unicancer will share de-identified individual data that underlie the results reported. A decision concerning the sharing of other study documents, including protocol and statistical analysis plan will be examined upon request.
Supporting Information: Study Protocol, SAP
Time Frame: The data shared will be limit to that required for independent mandated verification of the published results, the applicant will need authorization from Unicancer for personal access, and data will only be transferred after signing of a data access agreement.
Access Criteria: Unicancer will consider access to study data upon written detailed request sent to Unicancer, from 6 months until 5 years after publication of summary data.